CLINICAL TRIAL: NCT00332137
Title: Effects of Tolterodine, a Non-Specific Muscarinic Antagonist, on Gastrointestinal Transit in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1696-05
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Health
MeSH Terms: interventions — Tolterodine Tartrate

INTERVENTIONS:
Drug: Tolterodine

SUMMARY:
The muscarinic antagonist tolterodine is widely used treat urinary urge incontinence. Though acteylcholine is the primary excitatory neurotransmitter in the gastrointestinal tract, the phase III trials suggest that tolterodine infrequently causes constipation. Therefore, the objectives of this study are to assess if tolterodine affects the speed at which food travels through the stomach, intestines and colon (i.e., gastrointestinal and colonic transit) in healthy subjects.

DETAILED DESCRIPTION:
The specific aims of this study are to test the hypotheses that the non-specific muscarinic antagonist tolterodine will not:- i) delay colonic transit and the proximal colonic emptying rate; ii) delay gastric emptying; nor iii) delay small intestinal transit compared to placebo in healthy subjects.

ELIGIBILITY:
Age 18-70 years old. Absence of gastrointestinal symptoms as characterized by bowel symptoms questionnaire and absence of significant anxiety or depression characterized by a hospital anxiety and depression questionnaire.

Able to understand and willing to sign informed consent. Females who are nonpregnant, nonlactating, and willing to use a clinically approved methods of contraception two weeks prior to Day 0 until 1 week after the last dose of study medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2005-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Colonic transit (as measured by GC24)

SECONDARY OUTCOMES:
Colonic transit (GC48)
Ascending colon emptying t1/2
Colonic filling at 6 hours, i.e. a surrogate marker of small bowel transit time
Gastric emptying time (1, 2, 4 hours, thalf)
Average number of stools per day before and during treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States